CLINICAL TRIAL: NCT06456944
Title: Effect of Selected Rehabilitation Program on Pain, Function, and Plantar Fascia Thickness in Patients With Plantar Fasciitis
Brief Title: Effect of Selected Rehabilitation Program in Patients With Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohamed Ramadan Ibraheem Ramadan, principle investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mohamed PHD
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Plantar Fascitis; Plantar Fasciitis, Chronic; Heel Pain Syndrome
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Muscle Stretching Exercises; Ultrasonography; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: double blinded randomized controlled trial (participants blinded to the intervention and statistician blinded to group assignment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- selected rehabilitation program (Experimental): involves 24 patients and will be given the selected rehabilitation program involving (self-stretching exercise, mobilization of the ankle and subtalar, rigid tape and unilateral heel raising exercise 3 times per week for 8 weeks.
  Interventions: Other: stretching exercises; Other: rigid tape; Other: mobilization; Other: strengthening exercise
- traditional program (Experimental): involves 24 patients and will be given the traditional program involving (self-stretching exercise, mobilization of the ankle and subtalar, plantar fascial release and ultrasonic therapy 3 times per week for 8 weeks.
  Interventions: Other: stretching exercises; Device: ultrasound; Other: mobilization; Other: myofascial release

INTERVENTIONS:
Other: stretching exercises — stretching exercises of the plantar fascia, gastrocnemius and soleus
Device: ultrasound — therapeutic ultrasound upon the most painful point on the medial calcaneal tubercle. The parameters involved a pulsed mode (duty cycle 50%) using an intensity of 1.5 W/cm2 and a 1 MHz of frequency for 5 minutes
  Arms: traditional program
Other: rigid tape — low-dye tapping will be done to provide mechanical correction to plantar fascia and medial longitudinal arch
  Arms: selected rehabilitation program
Other: mobilization — mobilization techniques for the talocrural joint in weight bearing and non-bearing positions and subtalar joint
Other: myofascial release — deep tissue release of the plantar fascia and flexor hallucis longus in a stretched position of the plantar fascia
  Arms: traditional program
Other: strengthening exercise — strengthening exercise of the plantar intrinsic muscles using short foot exercise and strengthening of the Achilles tendon and windlass mechanism using unilateral heel raise exercises
  Arms: selected rehabilitation program

SUMMARY:
This study will be done to investigate the effect of the selected rehabilitation program for PF on plantar fascia thickness, clinical outcomes such as pain, foot function, dorsiflexion ROM and pressure pain threshold and alignment such as rearfoot eversion angle and foot posture index in patients with PF.

DETAILED DESCRIPTION:
Plantar fasciitis (PF), which constitutes approximately 15% of all foot disorders, is the most prevalent cause of heel pain. It is a long-term degenerative process that is impacted by subtalar pronation and pes planus. One million US patients saw primary care physicians with PF between 1995 and 2000. There is not enough data to determine the best physical therapy management techniques for individuals with heel pain, despite the existence of multiple successful treatment approaches. this study investigated at how a mechanically based rehabilitation program affected patients with PF in terms of foot alignment, plantar fascia thickness, pain, pressure pain threshold, ROM and foot function. The approach included strengthening the plantar intrinsic muscles of the foot, plantar fascia specific stretching and Achilles tendon stretching, and passively correcting the pathomechanics of the foot by low dye tapping and high load resistance exercise for Achilles tendon and windlass mechanism

ELIGIBILITY:
Inclusion Criteria:

* Plantar medial heel pain: most noticeable with initial steps after a period of inactivity, but also worse following prolonged weight-bearing
* Pain with palpation of the proximal insertion of the plantar fascia
* Positive windlass test
* flat foot posture utilizing the foot posture index
* age range from 40 to 60 years

Exclusion Criteria:

* tarsal tunnel syndrome
* atrophy of the fat pad.
* diabetic patients or patients with rheumatoid arthritis
* corticosteroid injection over the last sex months

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Assessing the change in pain intensity | At baseline and following 8 weeks
  VAS is typically composed of a 100 mm horizontal line attached to two opposed labels, the left end marked "no pain" and the right end marked "worst possible pain. Patients were marked a score on the scale by a vertical line that exactly refer to their pain

SECONDARY OUTCOMES:
Assessing the change in foot posture | At baseline and following 8 weeks
  using the foot posture index. It is a clinical measure of foot posture, either supinated or pronated, using 6 items for assessment of foot and scoring of each item from -2 to +2
Assessing the change in foot function | At baseline and following 8 weeks
  The Arabic version of the foot function index (FFI) is a widely used self-reporting measure used to assess the impact of foot pathology on pain, disability, and activity limitation. It is a reliable and sensitive outcome measure for patients with foot and ankle disorders. The FFI's subscale scores range from 0% to 100%, with higher scores indicating lower function and a poorer quality of life.
Assessing the change in plantar fascia thickness | At baseline and following 8 weeks
  using the ultrasound, participants were positioned in a prone position with relaxed arms and legs, and measurements were taken with the ankle joint in neutral or slightly dorsi-flexion. Electro-conductive gel was applied to the US transducer and plantar surface of foot before imaging. The transducer was placed longitudinally on the calcaneus surface to obtain a clear image of the plantar fascia.
Assessing the change in rear foot angle | At baseline and following 8 weeks
  using kinovea motion analysis software, the rearfoot (calcaneus) angle is measured as the angle between the bisection of the lower one-third of the leg and the bisection of the calcaneus. The MLA is classified as: normal arch 2-8°, low arch ≥ 8.1° and high arch ≤ 1.9.
Assessing the change in range of motion | At baseline and following 8 weeks
  The bubble inclinometer is used to measure the angle of the tibia relative to the floor during active ankle dorsiflexion, while the patient lunges forward with their heel on the ground and knee in line with the second toe.
Assessing the change in pressure pain threshold | At baseline and following 8 weeks
  the pressure algometer is utilized to measure the pressure pain threshold (PPT), The patient lay supine, in a relaxed position, with his feet hanging over the edge of the bed with no pressure on the heel. PPT is measured by laying the patient supine with feet hanging over the bed, without pressure on the heel. PPT is determined by applying pressure to the skin until the patient experiences pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ramadan Ibraheem, Assistant lecturer, Principal Investigator — Horus University
Locations (2):
- Egypt (2):
  - Outpatient clinic, Faculty of Physical Therapy, Horus University, Egypt, Damietta
  - out-patient clinic, Faculty of Physical Therapy, Horus university, Damietta